CLINICAL TRIAL: NCT06861790
Title: Obesity and Type 2 Diabetes: Bariatric Surgery Effects on Brain Function -Part 2 (WISE-2B Brain Study)
Brief Title: WISE-2B Brain Study (Weight Loss Intervention Surgical Effects on Brain Function)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: IRB202301845; R01DK099334 (NIH)
Record Dates: First submitted 2025-02-07; First posted 2025-03-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Diabetes; Weight Loss
Keywords: Weight loss and brain function; Effects of bariatric surgery on brain function; Reduced glucose insulin changes and brain function; tVNS intervention post-surgery
MeSH Terms: conditions — Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tVNS + anterior vagotomy (Experimental): This arm will receive transcutaneous vagus nerve stimulation and an anterior vagotomy during their bariatric surgery. Note a vagotomy is standard practice during bariatric surgery.
  Interventions: Behavioral: tVNS; Procedure: Anterior Vagotomy
- tVNS + complete vagotomy (Experimental): This arm will receive transcutaneous vagus nerve stimulation and a complete vagotomy during their bariatric surgery. Note a vagotomy is standard practice during bariatric surgery
  Interventions: Behavioral: tVNS; Procedure: Complete Vagotomy
- Sham + anterior vagotomy (Sham Comparator): This arm will not receive transcutaneous vagus nerve stimulation and will receive an anterior vagotomy during their bariatric surgery. Note a vagotomy is standard practice during bariatric surgery.
  Interventions: Procedure: Anterior Vagotomy
- Sham + complete vagotomy (Sham Comparator): This arm will not receive transcutaneous vagus nerve stimulation and will receive a complete vagotomy during their bariatric surgery. Note a vagotomy is standard practice during bariatric surgery.
  Interventions: Procedure: Complete Vagotomy

INTERVENTIONS:
Behavioral: tVNS — Though we will be utilizing a tVNS (Transcutaneous Vegus Nerve Stimulation) device this study is not a device study. The device being used is being done so under its approved usage. The intervention utilizes a non-invasive process to stimulate the Vagus nerve using very small electrical currents. This intervention is completed daily for one month.
  Arms: tVNS + anterior vagotomy; tVNS + complete vagotomy
Procedure: Complete Vagotomy — Participants will not be receiving bariatric surgery as an intervention of this study. Instead, the study will enroll patients already planning on undergoing the surgery. The surgeon will utilize one of two surgical approaches which will be observed in this study.
  Arms: Sham + complete vagotomy; tVNS + complete vagotomy
Procedure: Anterior Vagotomy — Participants will not be receiving bariatric surgery as an intervention of this study. Instead, the study will enroll patients already planning on undergoing the surgery. The surgeon will utilize one of two surgical approaches which will be observed in this study.
  Arms: Sham + anterior vagotomy; tVNS + anterior vagotomy

SUMMARY:
The goal of the study to understand the effects of weight loss and improvements in diabetes following bariatric surgery on brain function and thinking. This study will also examine whether non-invasive transcutaneous vagal nerve stimulation (tVNS) intervention initiated 30 days post-surgery improves brain function and thinking. The study does NOT cover any costs associated with bariatric surgery.

DETAILED DESCRIPTION:
There will be one group of study participants.

The group will (independently of this research study) have weight loss surgery to help them with weight loss.

All research participants in this group will be tested on thinking and memory processes at the start of the study, after 12 weeks, and again at 18 months. They will also undergo a non-invasive transcutaneous vagal nerve stimulation (tVNS) intervention days post-surgery, for 30 days at home with the device that is provided.

The group will have an MRI Brain Scan at each time-point to study the changes in the structure and function of the brain tissue.

Blood tests will be done to measure the sugar levels in the blood, and other proteins that may act as markers for disease.

ELIGIBILITY:
Inclusion Criteria:

* Between age: 20-75 yrs, English speaking, Physically mobile
* Body Mass Index (BMI) >35 kg before surgery
* Compatible of MRI Scanning
* Willing to give a small blood sample
* Capable of providing informed consent

Exclusion Criteria:

* Prior or current neurological disorder
* Major psychiatric disturbance
* Unstable medical conditions (cancer)
* MRI contraindications (claustrophobia, metal implants, waist/torso circumference)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Brain inflammation - MRS | 18 months
  Utilizing MRS the study seeks to understand changes in brain inflammation between the groups
Cognitive functioning - Global functioning score | 18 months
  Utilizing a battery of cognitive tests the study seeks to determine changes in cognitive functioning. This can be determined by computing the Global functioning score on the battery of measures.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Porges, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida - College of Public Health and Health Professions, Gainesville, Florida, United States